CLINICAL TRIAL: NCT02036710
Title: Location of Glucagon-Like Peptide (GLP)-1 Release
Brief Title: Location of GLP-1 Release
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1104M97972
Record Dates: First submitted 2014-01-10; First posted 2014-01-15 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Obesity
Keywords: GLP-1; PYY; Leptin; Duodenal Switch
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cecum: Food hydrolysate instilled into terminal cecum of patient undergoing open duodenal switch procedure. Blood samples were then obtained at baseline and at 0, 30, 60, 90, and 120 minutes for analysis of circulating GLP-1, PYY, and leptin.
- Ileum: Food hydrolysate instilled into terminal ileum of patient undergoing open duodenal switch procedure. Blood samples were then obtained at baseline and at 0, 30, 60, 90, and 120 minutes for analysis of circulating GLP-1, PYY, and leptin.

SUMMARY:
Background: Physicians do not have a unified, scientifically tested theory of causation for obesity and its comorbidities, nor do they have explanations for the mechanics of the metabolic/bariatric surgery procedures. Integral to proffered hypotheses are the actions of the hormones glucagon-like peptide (GLP-1), peptide YY (PYY), and leptin.

Study objective: To obtain blood levels of GLP-1, PYY, and leptin after stimulation of the terminal ileum and cecum by a static infusion of a food hydrolysate in morbidly obese patients undergoing a duodenal switch procedure.

Methods: Plasma levels of GLP-1, PYY, and leptin were obtained at 0, 30, 60, 90, and 120 minutes after instillation of 240 ml of a food hydrolysate into the ileum or cecum.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who was qualified and approved for bariatric surgery and elected to undergo open duodenal switch procedure.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population consisted of morbidly obese individuals who had decided to undergo open duodenal switch surgery
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2011-11; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
GLP-1 | 2 hours
  GLP- levels were measured at intervals over two hours after static bowel food hydrolysate was infused, in patients undergoing scheduled open duodenal switch procedure.
peptide YY (PYY) | 2 hours
  PYY levels were measured at intervals over two hours after static bowel food hydrolysate was infused, in patients undergoing scheduled open duodenal switch procedure.
Leptin | 2 hours
  Leptin levels were measured at intervals over two hours after static bowel food hydrolysate was infused, in patients undergoing scheduled open duodenal switch procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Buchwald, MD, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States